CLINICAL TRIAL: NCT06734078
Title: An Italian Multicenter Retrospective Observational Study to Assess the Clinical Characteristics and the Outcome of Patients With Relapsed or Refractory Diffuse Large B-cell Lymphoma Treated With Polatuzumab Vedotin Plus Rituximab (± Bendamustine) Under Named Patient Programme
Acronym: POSS
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: POSS
Record Dates: First submitted 2024-12-01; First posted 2024-12-16 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-12

CONDITIONS: DLBCL - Diffuse Large B Cell Lymphoma
Keywords: bendamustine; rituximab; polatuzumab vedotin
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Study designobservational, non-interventional, retrospective, multicenter study.

DETAILED DESCRIPTION:
The study focusing on information about the effectiveness and safety of polatuzumab vedotin plus rituximab (± bendamustine) in patients who received at least one dose of polatuzumab vedotin plus rituximab (± bendamustine) under the NPP (D.M. 7 Sep 2017) programme in the period between June 2019 and Feb 2020 in Italy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with relapsed or refractory DLBCL who received at least 1 dose of polatuzumab vedotin under the NPP (D.M. 7 Sep 2017) in the period between June 2019 and Feb 2020 in Italy.
2. Age ≥ 18 years at enrolment.
3. Written informed consent (if applicable).

Exclusion Criteria:

Patients with DLBCL treated with polatuzumab vedotin plus rituximab (± bendamustine) within a clinical trial context

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: DLBCL patients who received at least one dose of polatuzumab vedotin plus rituximab (± bendamustine) under the NPP (D.M. 7 Sep 2017) programme in the period between June 2019 and Feb 2020 in Italy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
overall response rate (ORR) | through study completion, an average of 2 years
  Effectiveness of polatuzumab vedotin plus rituximab (± bendamustine) in patients with relapsed or refractory DLBCL who have received at least one dose of polatuzumab vedotin plus rituximab (± bendamustine) under the NPP (D.M. 7 Sep 2017) in the period between June 2019 and Feb 2020 in Italy. This value is calculated as the sum of partial (PRR) and complete response rates (CRR) at end of treatment.

SECONDARY OUTCOMES:
Overall Survival (OS) | through study completion, an average of 2 years
  is the length of time from either the date of diagnosis or the start of treatment ...
Progression Free Survival (PFS) | through study completion, an average of 2 years
  the length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease
disease free survival (DFS) at 6 months | through study completion, an average of 2 years
  the time from random assignment to cancer recurrence or death from any cause.
frequency distribution of the causes of death | through study completion, an average of 2 years
  frequency
Mean treatment duration | through study completion, an average of 2 years
  Mean treatment duration
Incidence and type of adverse events and severe adverse events | through study completion, an average of 2 years
  Incidence
Proportion of patients with clinical disease progression | through study completion, an average of 2 years
  Proportion
Proportion of patients requiring one or more emergency department visits, hospitalizations, use of hematopoietic growth factors and antibiotics, and blood product transfusions | through study completion, an average of 2 years
  Proportion of patients with clinical disease progression
Best response rate (BRR) | through study completion, an average of 2 years
  Best response rate (BRR)
frequency distribution of the causes of treatment discontinuation | through study completion, an average of 2 years
  frequency distribution of the causes of treatment discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Pier Luigi Zinzani, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (9):
- Italy (9):
  - IRCCS Azienda Ospedaliero - Universitaria di Bologna, Bologna, Bologna
  - Casa Sollievo della Sofferenza - Reparto di Oncoematologia, San Giovanni Rotondo, Foggia
  - Azienda Ospedaliera Universitaria- Policlinico di Bari, Bari
  - Ospedale Oncologico Armando Businco, Cagliari
  - Ospedale Maggiore della Carità, Novara
  - Azienda Ospedaliera "Ospedali Riuniti Villa Sofia-Cervello", Palermo
  - CORE IRCCS Arcispedale Santa Maria Nuova, Reggio Emilia
  - Azienda Ospedaliera Santa Maria - SC di Oncoematologia, Terni
  - ULSS2 - Ospedale Civile Ca' Foncello - UO Ematologia, Treviso

IPD SHARING:
Plan to Share IPD: No